CLINICAL TRIAL: NCT03252392
Title: Does Autism Spectrum Disorder(ASD)Show Any Degree of Hearing Abnormalities? :A Preliminary Study
Brief Title: /Autism Spectrum Disorder(ASD)Hearing Abnormalities Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, weaam noaman mohamed, Principal invistigator, Assiut University
Other Study IDs: IRB17200055
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Autism Spectrum Disorder
Keywords: hearing and communication abnormalities
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with autism spectrum disorder: Children aged 3-12 years diagnosed to have mild to moderate autism spectrum disorder diagnosed by childhood autism spectrum disorder(CARS 35% or less)
- healthy non autistic age matched volunteers: children aged 3-12 years old never diagnosed to have autism spectrum disorder

SUMMARY:
Co morbidity rates of hearing loss in children with autism spectrum disorder are high and increasing.

Investigators are aiming to:

1. evaluate peripheral auditory and brain stem auditory function in children with autism spectrum disorder.
2. compare communication capabilities in autistic children having hearing abnormalities and autistic children with normal hearing.

DETAILED DESCRIPTION:
Full audiological evaluation is carried out to all participants including:

* pure tone and speech audiometry.
* Tympanometry and acoustic reflex threshold evaluation.
* Threshold auditory brain stem response for threshold determination in non co operative children not respond to pure tone,speech audiometry.
* Auditory brain stem response for neuro-otologic diagnosis.
* Transient evoked otoacoustic emissions in children proved to have normal hearing to detect minimal cochlear affection .
* Transient evoked otoacoustic emissions with contralateral masking. Communication evaluation is carried out to all participants using arabic language test(kotby et al,1995).

Investigators use childhood autism rating scale for (CARS) for diagnosis of autism spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-12 years diagnosed to have mild to moderate autism spectrum disorder diagnosed by childhood autism spectrum disorder(CARS 35% or less)

Exclusion Criteria:

* children with otitis media with effusion.
* Associated neurological deficit .

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children aged 3-12 years old attending phoniatric unit of assiut university from october 2017 t0 october 2020.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of autistic participants suffering from hearing abnormalities. | 3 years from october 2017 to october 2020
  Invistigators choose autistic children attending phoniatric unit in assiut university from october 2017 to october 2020 as they will go under complete audiological evaluation.

IPD SHARING:
Plan to Share IPD: Yes
De identified IPD for all primary and secondary out come measures will be made available.
Time Frame: 6 months after publication
Access Criteria: Data access requests will be reviewed by an external independent review panel,Requesters will be required to sign a data access agreement